CLINICAL TRIAL: NCT00116038
Title: A Comparison of Two Metal Surface Finishes (Proximal-Coated Titanium Surface Versus Mid-Coated Titanium Surface) on Femoral Components in Hip Arthroplasty
Brief Title: A Comparison of Two Metal Surface Finishes on Femoral Components in Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Kolding Sygehus (Other); Aarhus University Hospital (Other); Zimmer Biomet (Industry)
Responsible Party: Professor Kjeld Soballe, Aarhus University Hospital, Tage-Hansens Gade 2, 8000 Aarhus C
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030192
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis
Keywords: RSA; Osteoarthritis; Hip arthroplasty; DEXA
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Device: Femoral implant (Versys Fiber Metal Taper®)

SUMMARY:
The purpose of this study is to compare metal surface finishes (proximal-coated titanium surface versus mid-coated titanium surface) on femoral components in hip arthroplasty.

DETAILED DESCRIPTION:
In younger patients femoral components are most often implanted without the use of cement. A direct ingrowth of bone to the implant is crucial to the attainment of good results in those cases where cement is not employed.

The construction of a femoral implant, Versys Fiber Metal Taper®, by Zimmer includes a more extensive coating than previous femoral implants. The improved surface coating has been shown to provide these implants with better properties than those demonstrated by implants currently in general use.

Theoretically, the greater porous surface of mid-coated implants should:

* Encourage bone ingrowth through improved osteoconductive properties, however more extensive coating might change the loss of bone due to stress shielding later in time
* Improve anchorage of the implant due to the higher friction coefficient
* Result in fewer postoperative complaints measured with the Harris Hip Score and visual analog scale scores

The migration of femoral components will be evaluated by RSA, performing radiostereometric analyses at the Orthopaedic Center, Aarhus University Hospital. The follow-up RSA will be scheduled for week 1, as well as 3 months, 12 months and 2 years after surgery. Bone mineral density around the implanted femoral component will be examined by DEXA scan at week 1, as well as 1 year and 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary arthritis in the hip.
* Patients with sufficient bone density to allow uncemented implantation of a femoral component.
* Informed patient consent in writing.

Exclusion Criteria:

* Patients with neuromuscular or vascular disease in the affected leg.
* Patients found upon operation to be unsuited for uncemented acetabulum component.
* Patients who regularly take non-steroid anti-inflammatory drugs (NSAID) and cannot interrupt intake for the postoperative phase of the study.
* Patients with fracture sequelae.
* Female patients of childbearing capacity.
* Hip joint dysplasia.
* Sequelae to previous hip joint disorder in childhood.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
migration of femoral components evaluated by RSA

SECONDARY OUTCOMES:
BMD in the surrounding bone tissue of femoral components

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD., Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Orthopaedic Center, Aarhus University Hospital,, Aarhus, Denmark